CLINICAL TRIAL: NCT02363374
Title: Induction Chemotherapy Before or After Preoperative Chemoradiotherapy and Surgery for Locally Advanced Rectal Cancer: A Randomized Phase II Trial of the German Rectal Cancer Study Group
Brief Title: Induction Chemotherapy Before or After Preoperative Chemoradiotherapy and Surgery for Locally Advanced Rectal Cancer
Acronym: CAOAROAIO-12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. med. Claus Rödel (Other)
Collaborators: Johann Wolfgang Goethe University Hospital (Other); Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Claus Rödel, Prof. MD, Goethe University
Organization: Goethe University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAOAROAIO-12
Record Dates: First submitted 2015-02-03; First posted 2015-02-16 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Rectal Neoplasms; Rectal Cancer Stage II; Rectal Cancer Stage III
Keywords: Rectal cancer stage II; Rectal cancer stage III; Multimodality treatment of locally advanced rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Fluorouracil; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Chemotherapy -> Chemoradiotherapy (Active Comparator): Induction chemotherapy followed by chemoradiotherapy before surgery
  Interventions: Drug: Induction Chemotherapy arm A; Radiation: Radiation arm A; Procedure: Surgery
- Arm B: Chemoradiotherapy -> Chemotherapy (Experimental): Combined chemoradiotherapy followed by three cycles chemotherapy before surgery
  Interventions: Radiation: Radiation arm B; Drug: Chemotherapy arm B; Procedure: Surgery

INTERVENTIONS:
Drug: Induction Chemotherapy arm A — Patients receive three induction chemotherapy cycles, starting on day 1, 15 and 29, consisting of:
  Folinic acid: 400 mg/sqm, 2h-iv; Oxaliplatin: 100 mg/sqm, 2h-iv; 5-FU: 2400 mg/sqm, 46h-iv
  After a break of two weeks, radiotherapy starts combined with:
  5-FU: 250 mg/sqm per day, iv, on day 43-57, day 64-77 Oxaliplatin: 50 mg/sqm, day 43, 50, 64, and 71
  Other Names: all brands of Oxaliplatin are allowed; all brands of 5-fluorouracil (5-FU) are allowed; all brands of Folinic acid (FA) are allowed
  Arms: Arm A: Chemotherapy -> Chemoradiotherapy
Radiation: Radiation arm A — Radiotherapy: 28 x 1.8 Gy (total: 50.4 Gy), 5 fractions per week on day 43 -80
  Arms: Arm A: Chemotherapy -> Chemoradiotherapy
Radiation: Radiation arm B — Radiotherapy: 28 x 1.8 Gy (total: 50.4 Gy), 5 fractions per week on day 1- 38
  Arms: Arm B: Chemoradiotherapy -> Chemotherapy
Drug: Chemotherapy arm B — chemoradiotherapy is started according to the following schedule: 5-FU: 250 mg/sqm per day, iv, on day 1-14, day 22-35; Oxaliplatin: 50 mg/sqm, day 1, 8, 22, and 29.
  After a break of two and a half weeks, patients receive three chemotherapy cycles, starting on day 57, 71 and 85, consisting of:
  Folinic acid: 400 mg/sqm, 2h-iv; Oxaliplatin: 100 mg/sqm, 2h-iv; 5-FU: 2400 mg/sqm, 46h-iv
  Other Names: all brands of Oxaliplatin are allowed; all brands of 5-fluorouracil (5-FU) are allowed; all brands of Folinic acid (FA) are allowed
  Arms: Arm B: Chemoradiotherapy -> Chemotherapy
Procedure: Surgery — Surgery should be performed about 5 (arm B) or 6 (arm A) weeks after the last radiation or chemotherapy, i.e. around day 123

SUMMARY:
Preoperative 5-FU-based (5-fluorouracil) chemoradiotherapy (CRT), total mesorectal excision surgery, and 4 cycles of adjuvant 5-FU - as established by CAO/ARO/AIO-94 - is at present a standard of care for patients with locally advanced rectal cancer (UICC stage II and III). The phase III German CAO/ARO/AIO-04 trial showed, that the addition of oxaliplatin increased treatment efficacy in terms of early secondary efficacy endpoints (e.g. the pCR-rate). With a median follow-up of 50 months, the primary endpoint of this trial - disease free survival - was significantly improved in the oxaliplatin-containing treatment arm (3-year disease-free survival (DFS) 71.2% versus 75.9%, hazard ratio (HR) 0.79, 95% confidence interval (CI) 0.64-0.98, p=0.03). The hereby proposed randomized phase II trial CAO/ARO/AIO-12 aims at finding novel and innovative aspects of rectal cancer treatment, and will thus provide important information for defining the experimental arm in the upcoming large scale trial of the group. Compared to the current standard, in both study arms, the sequence of the three treatment modalities is modified, placing the chemotherapy block before surgery. The pre-operative sequence of chemotherapy -> chemoradiotherapy (arm A) has been shown to be feasible with no early tumor progression prior to definitive surgical resection in a small randomized phase II study from Spain. The sequence chemoradiotherapy -> chemotherapy (arm B) may be beneficial according to response kinetics considerations, and by maintaining a highly effective local treatment in the first place. Both approaches could avoid the problem of major compliance problems with post-operative adjuvant chemotherapy. CAO/ARO/AIO: German Rectal Cancer Study Group

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with histologically confirmed diagnosis of rectal cancer localised 0 - 12 cm from the anocutaneous line as measured by rigid rectoscopy (i.e. lower and middle third of the rectum)
* Staging requirements: High-resolution, thin-sliced (i.e. 3mm) magnetic resonance imaging (MRI) of the pelvis is the mandatory local staging procedure.
* MRI-defined inclusion criteria: presence of at least one of the following high risk conditions: any cT3 (clinical stage tumor-3) if the distal extent of the tumor is < 6 cm from anocutaneous line or cT3 in the middle third of the rectum (≥ 6-12 cm) with MRI evidence of extramural tumor spread into the mesorectal fat of more than 5 mm (>cT3b), or resectable cT4 tumors, or any clear cN+ (clinical staging nodes) based on MRI-criteria
* Trans-rectal endoscopic ultrasound (EUS) is additionally used when MRI is not definitive to exclude early cT1/T2 disease in the lower third of the rectum or early cT3a/b tumors in the middle third of the rectum.
* Spiral-CT of the abdomen and chest to exclude distant metastases.
* Aged at least 18 years. No upper age limit.
* WHO/ECOG (World Health Organisation/Eastern Cooperative Oncology Group) Performance Status ≤ 1
* Adequate haematological, hepatic, renal and metabolic function parameters: Leukocytes ≥ 3.000/mm^3, absolute neutrophil count (ANC) ≥ 1.500/mm^3, platelets ≥100.000/mm^3, Hb > 9 g/dl; Serum creatinine ≤ 1.5 x upper limit of normal; Bilirubin ≤ 2.0 mg/dl, serum glutamic-oxaloacetic transaminase (SGOT), serum glutamic-pyruvic transaminase (SGPT), and alkaline phosphatase (AP) ≤ 3 x upper limit of normal
* Informed consent of the patient

Exclusion Criteria:

* Lower border of the tumor localised more than 12 cm from the anocutaneous line as measured by rigid rectoscopy
* Distant metastases (to be excluded by CT scan of the thorax and abdomen)
* Prior antineoplastic therapy for rectal cancer
* Prior radiotherapy of the pelvic region
* Major surgery within the last 4 weeks prior to inclusion
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
* Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment (adequate: oral contraceptives, intrauterine device or barrier method in conjunction with spermicidal jelly).
* On-treatment participation in a clinical study in the period 30 days prior to inclusion
* Previous or current drug abuse
* Concomitant other antineoplastic therapy
* Serious concurrent diseases, including neurologic or psychiatric disorders (incl. dementia and uncontrolled seizures), active, uncontrolled infections, active, disseminated coagulation disorder
* Clinically significant cardiovascular disease in (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 6 months before enrolment
* Chronic diarrhea (> grade 1 according NCI CTCAE)
* Prior or concurrent malignancy ≤ 3 years prior to enrolment in study (Exception: non-melanoma skin cancer or cervical carcinoma FIGO (International Federation of Gynecology and Obstetrics) stage 0-1), if the patient is continuously disease-free
* Known allergic reactions on study medication
* Known dihydropyrimidine dehydrogenase deficiency
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule (these conditions should be discussed with the patient before registration in the trial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Number of patients with pathological complete response (pCR), i.e. ypT0N0. | 123 +30 days
  Efficacy (pCR) of induction chemotherapy followed by chemoradiotherapy, or the other way round, before surgery in patients with locally advanced rectal cancer.

SECONDARY OUTCOMES:
Safety of the respective combination sequences by Toxicity assessment according to NCI CTCAE V.4.0 | 5 years
Surgical morbidity | 123 +30 days
Surgical complications | 123 +30 days
Pathological staging | 123 +14 days
Tumor downstaging assessed by ypTNM (neoadjuvant pathological staging tumor nodes metastasis) findings in relation to initial cTNM (clinical stage tumor nodes metastasis) | 123 +14 days
Tumor regression grading according to Dworak | 123 +14 days
R0 resection rate; negative circumferential resection rate | 123 +14 days
Rate of sphincter-sparing surgery | 123 +14 days
Relapse-free survival (local / distant / overall) | 5 years
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Claus Rödel, Prof., MD, Principal Investigator — Head of Department of Radiation therapy and Oncology, Johann Wolfgang Goethe University Hospital
Locations (20):
- Germany (20):
  - University Clinic, Erlangen, Bavaria
  - RWTH Aachen, Aachen
  - University Clinic, Bochum
  - Clinic for Radiotherapy, Chemnitz
  - Diacura Clinic for Radiotherapy, Coburg
  - Internist Practice, Dresden
  - University Clinic, Dresden
  - University Clinic, Esslingen am Neckar
  - University Hospital Frankfurt Goethe University, Frankfurt
  - University Clinic, Freiburg im Breisgau
  - HELIOS Park-Klinikum Leipzig, Leipzig
  - University Clinic, Leipzig
  - University Clinic, Mannheim
  - Hospital Miria Hilf, Mönchengladbach
  - Pius Hospital Oldenburg, Oldenburg
  - University Clinic, Oldenburg
  - Hospital Barmherziger Brueder, Regensburg
  - University Clinic, Regensburg
  - University Clinic, Rostock
  - University Clinic, Würzburg

REFERENCES:
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Sauer R, Liersch T, Merkel S, Fietkau R, Hohenberger W, Hess C, Becker H, Raab HR, Villanueva MT, Witzigmann H, Wittekind C, Beissbarth T, Rodel C. Preoperative versus postoperative chemoradiotherapy for locally advanced rectal cancer: results of the German CAO/ARO/AIO-94 randomized phase III trial after a median follow-up of 11 years. J Clin Oncol. 2012 Jun 1;30(16):1926-33. doi: 10.1200/JCO.2011.40.1836. Epub 2012 Apr 23. PMID 22529255
- [Background] Rodel C, Liersch T, Becker H, Fietkau R, Hohenberger W, Hothorn T, Graeven U, Arnold D, Lang-Welzenbach M, Raab HR, Sulberg H, Wittekind C, Potapov S, Staib L, Hess C, Weigang-Kohler K, Grabenbauer GG, Hoffmanns H, Lindemann F, Schlenska-Lange A, Folprecht G, Sauer R; German Rectal Cancer Study Group. Preoperative chemoradiotherapy and postoperative chemotherapy with fluorouracil and oxaliplatin versus fluorouracil alone in locally advanced rectal cancer: initial results of the German CAO/ARO/AIO-04 randomised phase 3 trial. Lancet Oncol. 2012 Jul;13(7):679-87. doi: 10.1016/S1470-2045(12)70187-0. Epub 2012 May 23. PMID 22627104
- [Derived] Diefenhardt M, Fleischmann M, Martin D, Hofheinz RD, Piso P, Germer CT, Hambsch P, Grutzmann R, Kirste S, Schlenska-Lange A, Ghadimi M, Rodel C, Fokas E; German Rectal Cancer Study Group. Clinical outcome after total neoadjuvant treatment (CAO/ARO/AIO-12) versus intensified neoadjuvant and adjuvant treatment (CAO/ARO/AIO-04) a comparison between two multicenter randomized phase II/III trials. Radiother Oncol. 2023 Feb;179:109455. doi: 10.1016/j.radonc.2022.109455. Epub 2022 Dec 23. PMID 36572280
- [Derived] Fokas E, Schlenska-Lange A, Polat B, Klautke G, Grabenbauer GG, Fietkau R, Kuhnt T, Staib L, Brunner T, Grosu AL, Kirste S, Jacobasch L, Allgauer M, Flentje M, Germer CT, Grutzmann R, Hildebrandt G, Schwarzbach M, Bechstein WO, Sulberg H, Friede T, Gaedcke J, Ghadimi M, Hofheinz RD, Rodel C; German Rectal Cancer Study Group. Chemoradiotherapy Plus Induction or Consolidation Chemotherapy as Total Neoadjuvant Therapy for Patients With Locally Advanced Rectal Cancer: Long-term Results of the CAO/ARO/AIO-12 Randomized Clinical Trial. JAMA Oncol. 2022 Jan 1;8(1):e215445. doi: 10.1001/jamaoncol.2021.5445. Epub 2022 Jan 20. PMID 34792531
- See also: Related Info — https://www.kgu.de/einrichtungen/kliniken/zentrum-der-radiologie/strahlentherapie